CLINICAL TRIAL: NCT06509438
Title: Evaluating the Effectiveness and Safety of Embella (Deoxycholic Acid, Produced by Espad Pharmed Co.) for the Management of Submental Fat
Brief Title: Effectiveness and Safety Evaluation of Embella (Deoxycholic Acid, by Espad Pharmed Co.) in Management of Submental Fat
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Espad Pharmed (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: EMB.ESP.AF. IV.01
Record Dates: First submitted 2024-07-13; First posted 2024-07-19 (Actual); Results first posted 2025-09-19 (Actual); Last update posted 2025-09-19 (Actual); Status verified 2024-07

CONDITIONS: Submental Fullness

STUDY DESIGN:
Intervention Model Description: before/after clinical trial
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Embella (Deoxycholic acid, produced by Espad Pharmed Co.) (Experimental): The intervention included a minimum of one and a maximum of three treatment sessions, of 2 milliliters of Embella (Deoxycholic acid, produced by Espad Pharmed Co.) injectable solution containing 20 milligrams of deoxycholic acid per session, spaced at least 4 weeks apart.
  Interventions: Device: Embella (Deoxycholic acid, produced by Espad Pharmed Co.)

INTERVENTIONS:
Device: Embella (Deoxycholic acid, produced by Espad Pharmed Co.) — 2 milliliters of Embella injectable solution containing 20 milligrams of deoxycholic acid

SUMMARY:
Submental fat (SMF) is a factor affecting beauty that makes people feel uncomfortable about themselves. In 2015, deoxycholic acid with the brand name KYBELLA® was approved by the American FDA for treatment of submental fat. The purpose of this study is to evaluate the safety and effectiveness of deoxycholic acid injection with the brand name Embella®, manufactured by Espad Pharmed Company, for treatment of this condition.

Research Objectives

Primary objective:

Effectiveness and safety of Embella® in reducing submental fat

Secondary objective:

Effectiveness assessment of Embella® in improving SMF grading Effectiveness assessment of Embella® in reducing submental fat diameter

ELIGIBILITY:
Inclusion Criteria:

* Age between 18 and 65 years.
* Individuals with unwanted submental fat of any severity.
* Ability to comply with visit schedules and study procedures.
* Signed informed consent form and agreement to a 3-month follow-up.

Exclusion Criteria:

* Any previous intervention for the treatment of submental fat (SMF).
* Specific anatomical features or previous damage to the intervention site (e.g., scars, liposuction, swallowing difficulties, enlarged thyroid or lymph nodes) that could interfere with the assessment of intervention outcomes.
* Evidence of submental enlargement due to reasons other than SMF.
* History of dysphagia.
* Body mass index (BMI) > 30 kg/m².
* Individuals currently on a weight loss program.
* History of allergy to any components of the drug or local anesthetics.
* Presence of any inflammation, active infection, unhealed wounds, or skin lesions in the injection area.
* Use of any anticoagulants, NSAIDs, or any other medications that increase the risk of coagulation disorders within 7 days before injection.
* Unrealistic expectations.
* Pregnant or breastfeeding women.
* Individuals on sodium-restricted diets, such as those with uncontrolled hypertension.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2023-04-10 (Actual); Primary Completion 2024-01-01 (Actual); Study Completion 2024-01-01 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Center for Research and Training in Skin Diseases and Leprosy, Tehran, Iran

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Embella (Deoxycholic Acid, Produced by Espad Pharmed Co.)
Started | 20
Completed | 16
Not Completed | 4
Not completed — Adverse Event | 1
Not completed — Lost to Follow-up | 3

BASELINE CHARACTERISTICS:
Arm/Group | Embella (Deoxycholic Acid, Produced by Espad Pharmed Co.)
Number analyzed (Participants) | 20
Age, Continuous [Mean (Standard Deviation); unit: years] | 44.10 (11.35)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 17
  Male | 3
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  Iran | 20

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With A Minimum of One Grade Improvement in the Standard Submental Fat (SMF) Assessment Grading
Description: The scales are from 0 to 4, 0 indicating no localized submental fat and 4 indicating extreme submental convexity
Time Frame: Week 4 after the last injection, up to 12 weeks, and week 12 after the last injection, up to 20 weeks
Population: Analysis set includes only participants who had at least one post-baseline assessment of this outcome. One participant withdrew on Day 1 after the first injection due to an adverse event, and three participants were lost to follow-up by Week 12
Measure: Count of Participants; unit: Participants
Arm/Group | Embella (Deoxycholic Acid, Produced by Espad Pharmed Co.)
Number analyzed (Participants) | 19
Participants
  4 weeks after the last injection | 15
  12 weeks after the last injection: number analyzed (Participants) | 16
  12 weeks after the last injection | 10

2. Secondary Outcome: Measurement of Submental Fat Thickness
Description: Using calipers
Time Frame: Week 4 after the last injection, up to 12 weeks, and week 12 after the last injection, up to 20 weeks
Population: as for outcome 1
Measure: Median (Full Range); unit: Centimeters
Arm/Group | Embella (Deoxycholic Acid, Produced by Espad Pharmed Co.)
Number analyzed (Participants) | 20
Centimeters
  Baseline | 1.85 [1.60 to 2.70]
  4 weeks after the last injection: number analyzed (Participants) | 19
  4 weeks after the last injection | 1.40 [1.40 to 1.80]
  12 weeks after the last injection: number analyzed (Participants) | 16
  12 weeks after the last injection | 1.45 [1.40 to 1.90]
Statistical Analysis 1: Comparison: Embella (Deoxycholic Acid, Produced by Espad Pharmed Co.); Test type: Other — Compare 4 weeks after the last injection to baseline; p < 0.001, Wilcoxon (Mann-Whitney); Difference of medians = -0.45
Statistical Analysis 2: Comparison: Embella (Deoxycholic Acid, Produced by Espad Pharmed Co.); Test type: Other — Compare 12 weeks after the last injection to baseline; p < 0.001, Wilcoxon (Mann-Whitney); Difference of medians = -0.4

3. Secondary Outcome: Pain Intensity Was Assessed Using the VAS From 0 to 10
Description: Visual Analogue Scale (VAS): pain intensity scale where 0 indicates no pain and 10 indicates the maximum pain imaginable
Time Frame: Day 1, week 4 and week 8
Population: At each post-baseline visit the analysis includes only those participants who actually received an injection at that visit and provided a pain-after-injection assessment. The Day 0 (first) injection was mandatory for all enrolled participants, but all subsequent injections were optional 'touch-up' procedures given only when the investigator judged them necessary. Consequently, numbers analyzed are smaller at later time points.
Measure: Mean (Full Range); unit: units on a scale
Arm/Group | Embella (Deoxycholic Acid, Produced by Espad Pharmed Co.)
Number analyzed (Participants) | 20
units on a scale
  Day 1 | 5.1 [1 to 9]
  week 4: number analyzed (Participants) | 15
  week 4 | 3.9 [1 to 9]
  week 8: number analyzed (Participants) | 14
  week 8 | 3.0 [1 to 9]

4. Secondary Outcome: Subject Satisfaction Was Assessed Using the VAS From 0 to 10
Description: Visual Analogue Scale (VAS): satisfaction factor scale where 0 indicates complete dissatisfaction and 10 indicates maximum satisfaction
Time Frame: Week 4 after the last injection, up to 12 weeks, and week 12 after the last injection, up to 20 weeks
Population: as for outcome 1
Measure: Mean (Full Range); unit: units on a scale
Arm/Group | Embella (Deoxycholic Acid, Produced by Espad Pharmed Co.)
Number analyzed (Participants) | 19
units on a scale
  4 weeks after the last injection | 7.63 [1 to 10]
  12 weeks after the last injection: number analyzed (Participants) | 16
  12 weeks after the last injection | 7.43 [1 to 10]

5. Secondary Outcome: Number of Participants With Adverse Events Immediately After the Injections and During the Study Period
Description: Safety assessment: number of participants with adverse events
Time Frame: Immediately after all of the injections and at week 4 after the last injection, up to 12 weeks, and week 12 after the last injection, up to 20 weeks
Population: All subjects that received study treatment are included in the safety population.
Measure: Count of Participants; unit: Participants
Arm/Group | Embella (Deoxycholic Acid, Produced by Espad Pharmed Co.)
Number analyzed (Participants) | 20
Participants | 18

ADVERSE EVENTS:
Time Frame: Immediately after all of the injections and at week 4 after the last injection, up to 12 weeks, and week 12 after the last injection, up to 20 weeks
Arm/Group | Embella (Deoxycholic Acid, Produced by Espad Pharmed Co.)
All-Cause Mortality (participants affected / at risk) | 0/20
Serious Adverse Events (participants affected / at risk) | 0/20
Other Adverse Events (participants affected / at risk) | 18/20
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Embella (Deoxycholic Acid, Produced by Espad Pharmed Co.) (N=20)
Injection site tenderness (General disorders) | 13 (19)
Injection site numbness (General disorders) | 7 (9)
Injection site swelling (General disorders) | 4 (5)
Rigidity (General disorders) | 2 (3)
Globus sensation (General disorders) | 1 (2)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Skin laxity (Skin and subcutaneous tissue disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (2):
  • Study Protocol (2022-11-20): https://cdn.clinicaltrials.gov/large-docs/38/NCT06509438/Prot_000.pdf
  • Statistical Analysis Plan (2022-11-20): https://cdn.clinicaltrials.gov/large-docs/38/NCT06509438/SAP_001.pdf